CLINICAL TRIAL: NCT06767332
Title: EMDR for Fear of Cancer Recurrence in Patients with Familial Melanoma: a Waiting List Control Trial
Acronym: FAME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, schhinnen, dr. Chris (S.C.H.) Hinnen, Principal Investigator, Clinical Psychologist, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL79844.058.22
Record Dates: First submitted 2023-08-28; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Familial Melanoma; Fear of Cancer Recurrence; Eye Movement Desensitization and Reprocessing; Psychological Intervention
Keywords: EMDR; Fear of Cancer Recurrence; Familial Melanoma; Eye Movement Desensitization and Reprocessing; Psychological intervention; Anxiety; Psycho-oncology; FCR
MeSH Terms: conditions — Melanoma, Cutaneous Malignant; Anxiety Disorders | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Intervention Model Description: Randomised waiting-list controlled trial
Masking Description: Non-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Those assigned to the intervention condition will start EMDR treatment immediately after enrolment. The intervention will consist of an intake (90 min) and a maximum of 4 EMDR sessions (90 min each). After inclusion, baseline characteristic (sociodemographic and clinical variables) will be assessed. Moreover, before start EMDR treatment, after the last EMDR session and 2 weeks- and 3 months after ending EMDR treatment FCR and quality of life will be assessed.
  Interventions: Other: eye movement desensitization and reprocessing (EMDR)
- Waiting-list (No Intervention): Those assigned to the waiting-list will wait for 6 weeks. After these 6 weeks those assigned to the waiting list condition are able to receive the same treatment and the same assessment schedule when FCR is still present.

INTERVENTIONS:
Other: eye movement desensitization and reprocessing (EMDR) — EMDR is a psychological intervention that has historically been applied to the treatment of Post-Traumatic Stress Disorder (PTSD), but has since then been shown to be effective for a variety of anxiety disorders (e.g. fear of illness and specific phobia) (Logie & de Jongh, 2014) and somatic complaints such as post-operative pain, medically unexplained symptoms and seizure-related post-traumatic stress (Dautovic, de Roos, van Rood, Dommerholt, & Rodenburg, 2016; van Rood & de Roos, 2009; Maroufi, Zamani, Izadikhah, Marofi, & O'Connor, 2016).
  With more than 25 randomized clinical trials, EMDR has been established as an evidence-based intervention for PTSD and PTSD symptomatology including physical symptoms and fear of future catastrophes (Balkom van et al., 2013).
  Arms: Intervention

SUMMARY:
High fear of cancer recurrence (FCR) impacts patient's quality of life (QoL) and is prevalent among patients with familial melanoma. The main objective is to investigate whether EMDR is effective in treating high FCR in patients with familial melanoma. The study design is a non-blinded, randomized waiting-list controlled trial. Patients aged 18 years or older with familial melanoma can be included. Patients with high FCR will receive a maximum of 4, 90 minutes, EMDR-sessions. The main study parameter is the decrease and level of FCR measured with the Cancer Worry Scale (CWS). The secondary study parameter is quality of life, measured with the EORTC.

DETAILED DESCRIPTION:
There are an estimated 232100 cutaneous melanoma (CM) cases diagnosed and 55500 (24%) reported deaths worldwide annually. The incidence and mortality rates of CM vary per geographic location and the highest incidence rates are reported for Caucasian populations with fair skin. Approximately 10% of patients diagnosed with CM have a positive family history for this malignancy. CDKN2A gene (p16-leiden mutation) is the major melanoma susceptibility gene explaining approximately 35% of familial cases. Patients with hereditary melanoma due to a CDKN2A mutation have an estimated 70% risk of developing melanoma and a 20% risk of pancreatic cancer. Many patients with this type of melanoma develop melanoma at an earlier age than with non-familial melanoma and many develop multiple melanomas. Fear of cancer recurrence (FCR) has been found to be high (38%) among patients with CM and also among patients with familial melanoma. A large group of patients, about one third, indicate they need help with the uncertainty and threat of developing a new melanoma. While some amount of fear may be adaptive and bolster adequate healthcare behavior such as UV protection and skin examination, high levels of fear have a negative impact on patients quality of life and may lead to increased healthcare utilization. In most patients, fear of future catastrophes, such as illness recurrence, is based on past experiences.

Eye Movement Desensitization and Reprocessing (EMDR) is an intervention to desensitize both memories of past experiences as well as representations of future catastrophes. EMDR is an evidence-based and protocolized treatment for patients with Post Traumatic Stress Disorder (PTSD) and PTSD symptomatology including fear of future catastrophes. EMDR has been shown effective not only as treatment for PTSD but also for anxiety in the context of illness or medical situations. EMDR is already used in clinical practice as a treatment for FCR. Of late, is shown that EMDR-therapy is effective in decreasing FCR in patients with mammary- and colorectal carcinoma. In this study, with a replicated (n=8) single case experimental design, is found that EMDR had a large effect on high FCR and that 6 out of 8 patients went from high FCR to low FCR after EMDR. In the present study, the investigators will further investigate the effectiveness of EMDR in reducing FCR in patients with familial melanoma.

The investigators hypothesize that EMDR treatment will lead to a significant reduction of FCR in comparison to the waitinglist condition at the end of EMDR and at 2 weeks- and 3 months follow-up. The investigators hypothesize that EMDR treatment will improve the quality of life in comparison to the waiting list condition at the end of EMDR and at 2 weeks- and 3 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* a score of 16 or higher on the FCRI-NL-SF
* 18 years or older
* diagnosed with familial melanoma

Exclusion Criteria:

* insufficient knowledge of the Dutch language.
* acute psychiatric disease (psychosis, suicidal ideation)
* variable dosis of anxiolytics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Fear of Cancer Recurrence (FCR) | EMDR treatment takes approximately 4 weeks, waitinglist 6 weeks. CWS is filled in before randomisation (T0), after 4 weeks/at end of EMDR treatment (T1), after 6 weeks/2 weeks after ending EMDR treatment (T2) and 3 months after ending EMDR treatment (T3)
  FCR is measured with de Cancer Worry Scale (CWS). The CWS is able to detect high levels of FCR in a 6-item questionnaire (a 4 point Likert scale Ranging from 1 ("never") to 4 ("almost always"). Possible scores range from 6 to 24 with higher scores indicating more worry. The CWS is a much used and reliable and valid questionnaire to assess FCR in cancer survivors (Custers, et al., 2014).

SECONDARY OUTCOMES:
Quality of life (QoL) | EMDR treatment takes approximately 4 weeks. Waitinglist takes 6 weeks. EORTC-QLQ-C30 is filled in before randomisation (T0), after 6 weeks/2 weeks after ending EMDR treatment (T2) and at follow-up 3 months after ending EMDR treatment (T3).
  QoL is measured with the EORTC-QLQ-C30. The EORTC-QLQ-C30 has been developed for measuring health related quality of life in cancer patients (Aaronson, et al., 1993). The self-report questionnaire consists of 30 items of which 28 items are scored on a 4 points likert-scale and 2 items are scored on a 7 points likert-scale. The questionnaire contains functional and symptom subscales, and two items assessing general quality of life. The EORTC-QLQ-C30 is found to be reliable and valid for measuring the quality of life (Aaronson, et al., 1993, Groenvold, et al., 1997). The most recent version (3.0) has been tested in EORTC field studies (Bjordal, et al., 2000).

CONTACTS AND LOCATIONS:
Overall Officials: Chris Hinnen, Dr., Principal Investigator — Leiden University Medical Centre
Locations (2):
- Netherlands (2):
  - Leiden University Medical Center, Leiden, South Holland
  - Leiden University Medical Centre, Leiden, South Holland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hinnen C, Boonstra A, Kukutsch N, van Doorn R. Prevalence and indicators of fear of melanoma in patients with familial melanoma during surveillance. J Eur Acad Dermatol Venereol. 2021 Mar;35(3):e217-e218. doi: 10.1111/jdv.16939. Epub 2020 Oct 1. No abstract available. PMID 32936976
- [Background] Bruin J, van Rood YR, Peeters KCMJ, de Roos C, Tanious R, Portielje JEA, Gelderblom H, Hinnen SCH. Efficacy of eye movement desensitization and reprocessing therapy for fear of cancer recurrence among cancer survivors: a randomized single-case experimental design. Eur J Psychotraumatol. 2023;14(2):2203427. doi: 10.1080/20008066.2023.2203427. PMID 37144665
- [Background] Custers JA, van den Berg SW, van Laarhoven HW, Bleiker EM, Gielissen MF, Prins JB. The Cancer Worry Scale: detecting fear of recurrence in breast cancer survivors. Cancer Nurs. 2014 Jan-Feb;37(1):E44-50. doi: 10.1097/NCC.0b013e3182813a17. PMID 23448956
- [Background] Dautovic E, de Roos C, van Rood Y, Dommerholt A, Rodenburg R. Pediatric seizure-related posttraumatic stress and anxiety symptoms treated with EMDR: a case series. Eur J Psychotraumatol. 2016 Jul 4;7:30123. doi: 10.3402/ejpt.v7.30123. eCollection 2016. PMID 27387846
- [Background] Maroufi M, Zamani S, Izadikhah Z, Marofi M, O'Connor P. Investigating the effect of Eye Movement Desensitization and Reprocessing (EMDR) on postoperative pain intensity in adolescents undergoing surgery: a randomized controlled trial. J Adv Nurs. 2016 Sep;72(9):2207-17. doi: 10.1111/jan.12985. Epub 2016 May 1. PMID 27134066
- [Background] Shapiro F. The role of eye movement desensitization and reprocessing (EMDR) therapy in medicine: addressing the psychological and physical symptoms stemming from adverse life experiences. Perm J. 2014 Winter;18(1):71-7. doi: 10.7812/TPP/13-098. PMID 24626074
- [Background] Bell KJL, Mehta Y, Turner RM, Morton RL, Dieng M, Saw R, Guitera P, McCaffery K, Low D, Low C, Jenkins M, Irwig L, Webster AC. Fear of new or recurrent melanoma after treatment for localised melanoma. Psychooncology. 2017 Nov;26(11):1784-1791. doi: 10.1002/pon.4366. Epub 2017 Feb 2. PMID 28052599
- [Background] Champagne A, Ivers H, Savard J. Utilization of health care services in cancer patients with elevated fear of cancer recurrence. Psychooncology. 2018 Aug;27(8):1958-1964. doi: 10.1002/pon.4748. Epub 2018 Jun 1. PMID 29719072
- [Background] Fischbeck S, Imruck BH, Blettner M, Weyer V, Binder H, Zeissig SR, Emrich K, Friedrich-Mai P, Beutel ME. Psychosocial Care Needs of Melanoma Survivors: Are They Being Met? PLoS One. 2015 Aug 21;10(8):e0132754. doi: 10.1371/journal.pone.0132754. eCollection 2015. PMID 26296089
- [Background] Halk AB, Potjer TP, Kukutsch NA, Vasen HFA, Hes FJ, van Doorn R. Surveillance for familial melanoma: recommendations from a national centre of expertise. Br J Dermatol. 2019 Sep;181(3):594-596. doi: 10.1111/bjd.17767. Epub 2019 May 1. No abstract available. PMID 30742720
- [Background] Kasparian NA, McLoone JK, Butow PN. Psychological responses and coping strategies among patients with malignant melanoma: a systematic review of the literature. Arch Dermatol. 2009 Dec;145(12):1415-27. doi: 10.1001/archdermatol.2009.308. PMID 20026852
- [Background] Otto AK, Soriano EC, Siegel SD, LoSavio ST, Laurenceau JP. Assessing the relationship between fear of cancer recurrence and health care utilization in early-stage breast cancer survivors. J Cancer Surviv. 2018 Dec;12(6):775-785. doi: 10.1007/s11764-018-0714-8. Epub 2018 Oct 19. PMID 30341560
- [Background] Schadendorf D, van Akkooi ACJ, Berking C, Griewank KG, Gutzmer R, Hauschild A, Stang A, Roesch A, Ugurel S. Melanoma. Lancet. 2018 Sep 15;392(10151):971-984. doi: 10.1016/S0140-6736(18)31559-9. PMID 30238891
- [Background] Smith AB, Costa D, Galica J, Lebel S, Tauber N, van Helmondt SJ, Zachariae R. Spotlight on the Fear of Cancer Recurrence Inventory (FCRI). Psychol Res Behav Manag. 2020 Dec 21;13:1257-1268. doi: 10.2147/PRBM.S231577. eCollection 2020. PMID 33376421
- [Background] Wagner T, Augustin M, Blome C, Forschner A, Garbe C, Gutzmer R, Hauschild A, Heinzerling L, Livingstone E, Loquai C, Schadendorf D, Terheyden P, Mueller-Brenne T, Kahler KC. Fear of cancer progression in patients with stage IA malignant melanoma. Eur J Cancer Care (Engl). 2018 Sep;27(5):e12901. doi: 10.1111/ecc.12901. Epub 2018 Aug 20. PMID 30126009